CLINICAL TRIAL: NCT03538990
Title: Effect of Dietary Approaches to Stop Hypertension Eating Pattern on Cardiometabolic Markers in Advanced Heart Failure Patients
Brief Title: Effect of DASH Eating Pattern on Heart Failure Outcomes
Acronym: DASH HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Georgia (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Elisabeth Lilian Pia Sattler, Ph.D., B.S. Pharm, Assistant Professor, University of Georgia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005216
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Heart Failure NYHA Class III
Keywords: Nutrition; Dietary Approaches to Stop Hypertension; Cardiometabolic Outcomes; Pulmonary Artery Pressure; CardioMEMS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DASH Eating Pattern (Experimental): The DASH eating pattern meals prepared for study participants will strictly follow DASH meal planning guidelines published by National Heart, Lung, and Blood Institute of the National Institutes of Health. During the intervention phase of the study, all participants will exclusively consume prepared meals and provided beverages which will be delivered to participants' homes. Meals will be planned and prepared based on individual participant energy needs and dietary restrictions by a Registered Dietitian at the Georgia Clinical and Translational Science Alliance (CTSA) Bionutrition Unit located at Emory University.
  Interventions: Other: DASH Eating Pattern

INTERVENTIONS:
Other: DASH Eating Pattern — The DASH diet is a heart-healthy eating pattern that is focused on adequate consumption of fruits, vegetables, whole grains, low-fat dairy, fish, poultry, beans, nuts, and vegetables oils while emphasizing limited intake of foods containing saturated fat, such as fatty red meats, full-fat dairy products, and tropical oils, such as coconut, palm kernel, and palm oils, as well as sugar-sweetened beverages and sweets.

SUMMARY:
The objective of the study is to examine the effect of nutritional intake on cardiometabolic, inflammation, and physical function markers in advanced heart failure patients using a one-group pre-post test design feeding trial. Effects on hemodynamic markers will be assessed in a subsample of patients with implanted hemodynamic monitoring devices (CardioMEMS). The pre-test condition is represented by participants' self-selected diet, and the post-test condition is represented by a prescribed Dietary Approaches to Stop Hypertension (DASH) diet.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age
2. English language literacy
3. Diagnosis of HF ≥ 3 months
4. Diagnosis of NYHA Class III HF (historical assessment)
5. Subjects must be stable on HF medication regimen for one month prior to study entry
6. At least 1 HF hospitalization within 24 months of enrollment
7. BNP >200 pg/ml

Exclusion Criteria:

1. Subjects who have had an unplanned HF-related hospitalization within 2 months of enrollment
2. Subjects with a Glomerular Filtration Rate (GFR) <25 ml/min who are nonresponsive to diuretic therapy or who are on chronic renal dialysis
3. Subjects likely to undergo heart transplantation within 2 months of enrollment
4. Subjects with severe conditions limiting 6-month survival
5. Unavailability during scheduled data collection points
6. Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiometabolic Marker Levels between Calibration and DASH Diet Intervention Phase | Baseline, week 3, week 6
  Change of the following cardiometabolic marker values will be calculated between calibration and intervention phase using repeated measures analysis methods (3 time points over the course of 6 weeks: baseline, mid-point, post-DASH intervention): fasting lipid panel, hemoglobin A1c, basic metabolic panel (sodium, potassium, chloride, carbon dioxide (CO2), blood urea nitrogen, creatinine, and glucose), B-type natriuretic peptide (BNP), N terminal proBNP, troponin 1, mid-regional pro-adrenomedullin (MR-proADM), soluble somatostatin receptor 2 (sST2).

SECONDARY OUTCOMES:
Change in Functional Exercise Capacity between Calibration and DASH Diet Intervention Phase | Baseline, week 3, week 6
  We will compare the change in functional exercise capacity using the American Thoracic Society 6-minute walk test between calibration and intervention phase using repeated measures analysis methods (3 time points over the course of 6 weeks: baseline, mid-point, post-DASH intervention).

OTHER OUTCOMES:
Change in Inflammation Marker Levels between Calibration and DASH Diet Intervention Phase | Baseline, week 3, week 6
  We will compare the change of the following inflammation marker values between calibration and intervention phase using repeated measures analysis methods (3 time points over the course of 6 weeks: baseline, mid-point, post-DASH intervention): interleukin (IL)-1a, IL-1b, IL-6, and tumor necrosis factor alpha (TNF-a).
Change in Hemodynamic Marker Levels between Calibration and DASH Diet Intervention Phase | week 1-3, week 3-6
  Change in mean hemodynamic marker levels will be calculated by comparing mean values from the calibration (week 1-3) and intervention phase (week 3-6). All patients will be instructed to take daily pulmonary artery pressure home readings for the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth L Sattler, PhD, BSPharm, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia Clinical and Translational Research Unit, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided